CLINICAL TRIAL: NCT01949025
Title: Prevention of Serious Adverse Events in Acute Care Hospitals by Afferent Limb and Response Method Intervention - the ALARM Intervention Study.
Acronym: ALARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Belgian Federal Public Service, Food Chain Safety and Environment (Other Government)
Responsible Party: Principal Investigator, Filip Haegdorens, RN, MScN, PhD Candidate, Universiteit Antwerpen
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: ALARM1
Record Dates: First submitted 2013-09-17; First posted 2013-09-24 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Unexpected Hospital Mortality; Death, Sudden, Cardiac; Unplanned Intensive Care Unit Admission
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALARM intervention (Experimental): The training of nursing and medical staff about the observation, detection, assessment and communication of deteriorating and critically ill patients and the introduction of a standardized observation and communication protocol on medical and surgical wards.
  Interventions: Other: ALARM intervention
- Control group (No Intervention)

INTERVENTIONS:
Other: ALARM intervention — The training of nursing and medical staff about the observation, detection, assessment and communication of deteriorating and critically ill patients and the introduction of a standardized observation and communication protocol on medical and surgical wards.
  Arms: ALARM intervention

SUMMARY:
1. Summary

   Growing evidence suggests that a significant proportion of in-hospital patient deaths occur after serious adverse events (SAE's). Concerns have been raised that too often patients' acute deteriorations, particularly on surgical and medical wards outside critical care settings, are identified too late and corrective actions taken too slowly. Many initiatives have been taken to prevent unexpected death by timely recognition, intervention and resuscitation efforts such as Rapid Response Systems (RRS's). RRS's have been introduced with the intention to prevent SAE's and to improve patient outcome by facilitating early detection of warning signs for clinical deterioration. These systems have four components (1) an afferent limb for detection and response triggering, (2) an efferent limb with medical or nursing response to prevent deterioration (3) a process improvement limb and (4) a governance and administrative structure. It remains uncertain which elements of RRS's contribute most to patient outcomes such as unplanned (re-) admission to the intensive care unit, shock, cardiac arrest and unexpected death. In addition, previous studies found that nurse observation, assessment and communication (afferent limb) are crucial to achieve better patient outcomes, but how to achieve afferent limb sustainability in hospitals is not clear.

   A previous study investigated 23 hospitals in Flanders (Belgium) about how nurses observe, assess, detect and communicate deteriorating and critical patients in surgical, medical and geriatric wards. Wide variation between hospitals was identified about critical patient intervention procedures, strategies and Do Not Attempt Resuscitation (DNAR) orders as well as between nurses about the use and knowledge of critical vital signs and call criteria for physician clinical advice and support. Nurses of hospitals with structured observation and communication protocols were better informed and perceived their communication and collaboration with physicians more favorable in compared to other hospitals. Based on these results conclusions and recommendations for further initiatives were formulated. The proposed Afferent Limb and Response Method intervention study will implement these recommendations guided by a robust scientific research approach to offer evidence to the nursing and medical practice community.

   The aim of this study is to evaluate the effect of the Afferent Limb Ascertainment and Response Method intervention or ALARM intervention in medical and surgical nursing wards of acute care hospitals on the prevention of SAE's such as in-hospital unexpected death, unplanned ICU-admission and cardiac arrest.
2. Study hypothesis

Optimizing and supporting the process of observation, use and interpretation of vital signs, detection, assessment, escalation and communication with a higher level of care in deteriorating patients can prevent serious adverse events (in-hospital unexpected death, unplanned ICU admission and cardiac arrest) in acute care hospitals.

DETAILED DESCRIPTION:
- What does the study involve?

The study is based on the application of training and tools: the training of nursing and medical staff about the observation, detection, assessment and communication of deteriorating and critically ill patients and the introduction of a standardized observation and communication protocol on medical and surgical wards (tools). A training team will offer standardized training sessions.

- When does the study take place?

From October 1st 2013 till September 30th 2015.

- Where does the study take place?

Belgium.

- What are the risks to participants?

Patients will not be exposed to complementary risks if they partake in this study. No additional investigations will be performed for the purpose of this study since the aim of the intervention is to optimize existing processes that are already used in a hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the partaking wards during the study period (October 1st 2013 - September 30th 2015)

Exclusion Criteria:

* Age: ≤ 16

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69656 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
In-hospital unexpected death | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Unplanned ICU admission | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Cardiac arrest | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Filip Haegdorens, RN, MScN, PhD Candidate, Principal Investigator — Universiteit Antwerpen; Peter Van Bogaert, RN, MA, PhD, Study Chair — Universiteit Antwerpen; Koenraad G. Monsieurs, MD, PhD, Study Chair — Universiteit Antwerpen; Koen De Meester, RN, MScN, PhD, Study Chair — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Wilrijk, Antwerp, Belgium

REFERENCES:
- [Background] De Meester K, Haegdorens F, Monsieurs KG, Verpooten GA, Holvoet A, Van Bogaert P. Six-day postoperative impact of a standardized nurse observation and escalation protocol: a preintervention and postintervention study. J Crit Care. 2013 Dec;28(6):1068-74. doi: 10.1016/j.jcrc.2013.07.061. Epub 2013 Sep 6. PMID 24011975
- [Derived] Haegdorens F, Monsieurs KG, De Meester K, Van Bogaert P. An intervention including the national early warning score improves patient monitoring practice and reduces mortality: A cluster randomized controlled trial. J Adv Nurs. 2019 Sep;75(9):1996-2005. doi: 10.1111/jan.14034. Epub 2019 Jun 6. PMID 31012124
- See also: Related Info — http://www.alarmstudy.be